CLINICAL TRIAL: NCT05358769
Title: Randomized Clinical Trial to Assess the Effectiveness of Incoxil Food Supplement and Pelvic Floor Muscle Training in Women With Stress Dominant Urinary Incontinence.
Brief Title: A Study of Incoxil Food Supplement in Female Patients With Stress Dominant Urinary Incontinence.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FEMPHARMA Kft. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2022INCOXIL
Record Dates: First submitted 2022-04-28; First posted 2022-05-03 (Actual); Last update posted 2023-02-15 (Actual); Status verified 2023-02

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incoxil supplement group (Experimental): Incoxil supplement-group: receive daily oral Incoxil supplementation and perform pelvic floor muscle exercise (PFME) for 6 weeks.
  Interventions: Dietary Supplement: Incoxil food supplement and pelvic floor muscle exercise
- Control group (Active Comparator): Control group: receive placebo oral daily supplementation and perform pelvic floor muscle exercise (PFME) for 6 weeks.
  Interventions: Other: Pelvic floor muscle exercise

INTERVENTIONS:
Dietary Supplement: Incoxil food supplement and pelvic floor muscle exercise — Incoxil supplement group receives standardized written and verbal instructions on how to perform PFME and are asked to perform the pelvic floor muscle exercises 3 times per day, with 15 repetitions per set, daily for 6 weeks. Women perform PFME at an intensity of at least 65-75% of one repetition maximum. (Repetition maximum load is the maximum weight or force an individual can exert in a single lift.) In addition participants receive Incoxil food supplement and take the supplement once a day.
  Incoxil composition: creatine, l-leucine, zinc, calcium and magnesium. Incoxil is specifically designed to contain ingredients that help strengthen muscles during regular resistance training of moderate intensity.
  Arms: Incoxil supplement group
Other: Pelvic floor muscle exercise — Group receives standardized written and verbal instructions on how to perform PFME and are asked to perform the pelvic floor muscle exercises 3 times per day, with 15 repetitions per set, daily for 6 weeks. Women perform PFME at an intensity of at least 65-75% of one repetition maximum. (Repetition maximum load is the maximum weight or force an individual can exert in a single lift.) In addition participants receive placebo food supplement to take once a day.
  Arms: Control group

SUMMARY:
The purpose of this study is compare the effectiveness of Incoxil food supplement and pelvic floor muscle training with pelvic floor muscle training alone in the treatment of women with stress dominant urinary incontinence.

DETAILED DESCRIPTION:
Pelvic floor muscle training (PFMT) is the first line therapy recommended for the treatment of stress urinary incontinence. The study aims to investigate how poor pelvic floor muscle function can be strengthened by performing pelvic floor exercise and using a special dietary supplement at the same time, and if stress urinary incontinence can be improved more effectively than by performing pelvic floor exercise alone.

The study aims to compare the clinical improvement in the symptoms of stress urinary incontinence in women who do pelvic floor muscle training exercise (PFMT) or who do PFMT exercise and use a dietary supplement. Incoxil dietary supplement contains ingredients that are specifically designed to help strengthen muscles (creatine, l-leucine, zinc, calcium and magnesium).

The randomized controlled clinical trial is proposed involving 34 women diagnosed with stress dominant urinary incontinence and randomized into two groups: 1) treatment with Incoxil dietary supplement and PFMT; 2) treatment with placebo dietary supplement and PFMT. All women will perform PFMT daily and women in group 1 take Incoxil every day, while women in the control group will take daily placebo dietary supplement for 6 weeks.

At baseline assessment, patients shall undergo anamnesis, general gynecological exam, assessments of the pelvic floor based on the modified Oxford scale, the presence of prolapse using the Pelvic Organ Prolapse Quantification (POP-Q) system, pelvic muscle contraction will be measured using a pelvic Perineometer and Vaginal Tactile Imaging will be used for evaluation of vaginal and pelvic floor conditions. We also assess the general health of the vagina with Vaginal Health Index scores. Participants shall complete UDI-6, PGI-S/I and IIQ-7 questionnaires.

After 6 weeks treatment the same assessments will be done to compare treatment and control group results.

ELIGIBILITY:
Inclusion Criteria:

* stress UI or stress-dominant mixed UI (stress percent score more than urge percent score)

Exclusion Criteria:

* pregnancy or less than 12-month postpartum
* more than three vaginal deliveries or any prior operative delivery
* self-reported symptoms of pelvic organ prolapse or POP-Q stage >2
* history of supervised PFMT within 12 months
* current medications for UI
* known zinc or copper deficiency or sensitivity
* connective tissue disease

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2022-04-27 (Actual); Primary Completion 2022-09-09 (Actual); Study Completion 2022-09-09 (Actual)

PRIMARY OUTCOMES:
UDI-6 score | 6 weeks
  Comparison of Urogenital Distress Inventory-6 (UDI-6) questionnaire final scores before and after treatment in the two arms.

SECONDARY OUTCOMES:
Incontinence Impact Questionnaire (IIQ-7) score | 6 weeks
  Comparison of Incontinence Impact Questionnaire (IIQ-7) questionnaire final scores before and after treatment in the two arms.
Patient's Global Impression of Severity (PGI-S) | 6 weeks
  Comparison of Patient's Global Impression of Severity (PGI-S) questionnaire final scores before and after treatment in the two arms.
Patient's Global Impression of Improvement (PGI-I) | 6 weeks
  Patients will be asked answer the PGI-I questionnaire after the 6 week course of therapy.
Vaginal Tactile Imager (VTI) score | 6 weeks
  VTI is used for evaluation of vaginal and pelvic floor conditions at week 0 and week 6, before and after treatment. VTI allows assessment of tissue elasticity, pelvic floor support and function.
Vaginal squeeze pressure | 6 weeks
  Pelvic muscle contraction will be measured at week 0 and week 6 using a pelvic perineometer to assess any improvement in pelvic muscle strength.

CONTACTS AND LOCATIONS:
Overall Officials: Bence Kozma, MD PhD, Principal Investigator — Dr. Secret Private Clinic Debrecen Hungary
Locations (1):
- Dr. Secret Private Clinic, Debrecen, HB, Hungary

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Takacs P, Pakozdy K, Koroknai E, Erdodi B, Krasznai Z, Kozma B. A randomized controlled pilot trial to assess the effectiveness of a specially formulated food supplement and pelvic floor muscle training in women with stress-predominant urinary incontinence. BMC Womens Health. 2023 Jun 20;23(1):321. doi: 10.1186/s12905-023-02476-z. PMID 37340306